CLINICAL TRIAL: NCT00378703
Title: The BeST Trial: A Randomized Phase II Study of VEGF, RAF Kinase, and mTOR Combination Targeted Therapy (CTT) With Bevacizumab, Sorafenib, and Temsirolimus in Advanced Renal Cell Carcinoma
Brief Title: Bevacizumab, Sorafenib Tosylate, and Temsirolimus in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00533; NCI-2009-00533 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E2804; CDR0000499788; E2804 (Other: ECOG-ACRIN Cancer Research Group); E2804 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2015-05-05 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Sorafenib; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (bevacizumab) (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm B (bevacizumab and temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 and bevacizumab as in Arm A.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus
- Arm C (bevacizumab and sorafenib tosylate) (Experimental): Patients receive bevacizumab as in Arm A and sorafenib tosylate PO BID on days 1-5, 8-12, 15-19, and 22-26.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sorafenib Tosylate
- Arm D (sorafenib tosylate and temsirolimus) (Experimental): Patients receive sorafenib tosylate PO BID on days 1-28 and temsirolimus as in Arm B.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sorafenib Tosylate; Drug: Temsirolimus

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm A (bevacizumab); Arm B (bevacizumab and temsirolimus); Arm C (bevacizumab and sorafenib tosylate)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm C (bevacizumab and sorafenib tosylate); Arm D (sorafenib tosylate and temsirolimus)
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm B (bevacizumab and temsirolimus); Arm D (sorafenib tosylate and temsirolimus)

SUMMARY:
This randomized phase II trial studies different combinations of bevacizumab, temsirolimus, and sorafenib tosylate to see how well they work compared with bevacizumab alone in treating patients with kidney cancer that has spread to other places in the body. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab and sorafenib tosylate may stop the growth of tumor cells by blocking blood flow to the tumor. Temsirolimus and sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving different combinations of bevacizumab, sorafenib tosylate, and temsirolimus may be more effective than bevacizumab alone in treating metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess progression-free survival on each arm of combination targeted therapy (CTT) compared to that of bevacizumab alone.

SECONDARY OBJECTIVES:

I. To assess the significance of changes in tumor size over early time points as a predictor of progression-free survival (PFS).

II. To quantify the number and percent of patients who have stable disease at 6 months of therapy (failure to progress) in each treatment arm of CTT in patients with metastatic renal cell carcinoma (RCC).

III. To evaluate the safety of each treatment arm of combination targeted therapy (CTT) in patients with metastatic RCC.

IV. To assess overall survival in each arm of the study. V. To assess the objective response rate in each treatment arm of CTT in patients with metastatic RCC.

VI. To assess pathology, angiogenesis histology and to assess activation status of mitogen activated protein (MAP) kinase and vascular endothelial growth factor receptor 2 (VEGFR2) pathways and relate to clinical outcome.

TERTIARY OBJECTIVES:

I. To analyze the pharmacokinetic and pharmacogenetic properties of sorafenib (sorafenib tosylate) including angiogenesis, monooxygenases polymorphisms and multi-drug resistance (MDR).

II. To relate changes in tumor perfusion and vascular permeability on serial dynamic contrast-enhanced magnetic resonance imaging (MRI) to clinical outcome and radiologic regression detected by other standard methods.

III. To assess the potential of dynamic contrast-enhanced (DCE)-MRI imaging as a biomarker for response to therapy and/or as a prognostic indicator of disease progression.

IV. To assess site readiness and ability in acquiring DCE-MRI data. V. To determine the relationship between tumor and blood biomarkers and clinical outcomes of patients treated with the combination of targeted agents.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM A: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15.

ARM B: Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 and bevacizumab as in Arm A.

ARM C: Patients receive bevacizumab as in Arm A and sorafenib tosylate orally (PO) twice daily (BID) on days 1-5, 8-12, 15-19, and 22-26.

ARM D: Patients receive sorafenib tosylate PO BID on days 1-28 and temsirolimus as in Arm B.

In all arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be required to have the clear cell variant of renal cell carcinoma with less than 25% of any other histology (including, but not limited to, papillary or chromophobe or oncocytic); there must be histologic confirmation by treating center of either primary or metastatic lesion
* Patients will be required to have measurable metastatic disease that is not curable by standard radiation therapy or surgery; all sites must be assessed within 4 weeks prior to study entry
* Previous nephrectomy is required with the following exceptions:

  * Primary tumor =< 5 cm, or
  * Extensive liver (> 30% of liver parenchymal) or multiple (> 5) bone metastases, making nephrectomy a clinically questionable procedure
  * Unresectable primary tumor due to invasion into adjacent organs or encasing the aorta or vena cava
* No prior cytotoxic chemotherapy; a maximum of one prior regimen of either vaccine or cytokine-based immunotherapy disease is permitted
* No prior anti-angiogenic therapy including, but not limited to, SU11248, ZD6474 or VEGF Trap; no prior therapy with bevacizumab, mammalian target of rapamycin (mTOR) inhibitors (including, but not limited to, temsirolimus), or sorafenib will be allowed; thalidomide or interferon alpha (IFNalpha) are allowed either for adjuvant therapy or stage IV disease
* No immunotherapy within 4 weeks of randomization; toxicities from immunotherapy must have resolved and a minimum of two weeks must pass prior to enrollment
* Prior radiation therapy is permitted, but toxicities from radiation must have resolved and a minimum of 2 weeks must pass prior to randomization
* No history or clinical evidence of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastasis, or history of stroke within the past 48 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of greater than 12 weeks
* Hemoglobin (Hgb) >= 9.0 g/dL (transfusions allowed prior to enrollment)
* White blood count (WBC) >= 3,000/mm^3
* Absolute granulocyte count (AGC) >= 1,200/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or serum creatinine clearance (CrCl) >= 55 ml/min
* Total bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (or =< 5.0 x ULN in the presence of liver metastases)
* International normalized ratio (INR) =< 1.5
* Activated partial thromboplastin time (aPTT) within normal limits
* Fasting cholesterol < 350 mg/dL (9.0 mmol/L)
* Fasting triglycerides < 400 mg/dL (4.56 mmol/L)
* Patients must not have other current malignancies, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast; patients with other malignancies are eligible if they have been continuously disease-free for >= 5 years prior to the time of randomization
* No history of allergic reactions attributed to Chinese hamster ovary cell products, other recombinant human antibodies, or compounds of similar chemical or biologic composition to sorafenib, temsirolimus or bevacizumab
* No history of bleeding diathesis or coagulopathy
* Any condition that impairs patient's ability to swallow pills will make patient ineligible
* No major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomization
* No anticipated need for major surgery during the course of the study
* No current or recent (within 4 weeks of enrollment) use of full-dose of anticoagulants or thrombolytic agents (except as required to maintain patency of preexisting or permanent indwelling IV catheters, for those patients receiving warfarin, INR must be =< 1.5)
* No clinically significant cardiovascular disease, defined as one of the following:

  * Patients with uncontrolled hypertension (blood pressure > 150/100 mm/Hg at the time of enrollment); patients with hypertension and blood pressure =< 150/100 mm/Hg on stable antihypertensive regimen are eligible
  * Myocardial infarction or unstable angina < 24 weeks prior to registration
  * New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris
  * Grade II or greater peripheral vascular disease
* No serious, non-healing wound, ulcer, or bone fracture
* No significant proteinuria at baseline; urine protein must be screened within 2 weeks prior to randomization by urine analysis for urine protein creatinine (UPC) ratio; if UPC ratio is > 0.5, 24-hour urine protein is to be obtained and the level must be < 1000 mg for patient enrollment

  * NOTE: UPC ratio of spot urine is an estimation of the 24 urine protein excretion; a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics on day 0 or psychiatric illness/social situations that would limit compliance with study requirements
* Patients currently taking any of the following cytochrome P450 enzyme-inducing drugs are ineligible:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Rifampin
* Pregnant and breastfeeding women are excluded from the study; breastfeeding should be discontinued while receiving therapy; patients must have pregnancy test within 7 days prior to patient randomization if woman is of child-bearing capacity
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2007-09-14 (Actual); Primary Completion 2014-02-07 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Flaherty, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (559):
- United States (558):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - AMG Oncology - Naperville, Naperville, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Horizon Oncology Research LLC, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology-Austin North, Austin, Texas
  - Texas Oncology Seton Northwest, Austin, Texas
  - The Center for Cancer and Blood Disorders-Burleson, Burleson, Texas
  - Texas Oncology-Cedar Park, Cedar Park, Texas
  - The Center for Cancer and Blood Disorders-Cleburne, Cleburne, Texas
  - The Center for Cancer and Blood Disorders-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - The Center for Cancer and Blood Disorders-Mineral Wells, Mineral Wells, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Texas Oncology- San Marcos, San Marcos, Texas
  - The Center for Cancer and Blood Disorders-Weatherford, Weatherford, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Fox Valley Hematology and Oncology SC-Appleton, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - UW Health Oncology-One South Park, Madison, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

REFERENCES:
- [Derived] Flaherty KT, Manola JB, Pins M, McDermott DF, Atkins MB, Dutcher JJ, George DJ, Margolin KA, DiPaola RS. BEST: A Randomized Phase II Study of Vascular Endothelial Growth Factor, RAF Kinase, and Mammalian Target of Rapamycin Combination Targeted Therapy With Bevacizumab, Sorafenib, and Temsirolimus in Advanced Renal Cell Carcinoma--A Trial of the ECOG-ACRIN Cancer Research Group (E2804). J Clin Oncol. 2015 Jul 20;33(21):2384-91. doi: 10.1200/JCO.2015.60.9727. Epub 2015 Jun 15. PMID 26077237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between September 14, 2007 and December 10, 2010 with a final accrual of 361 patients.
Groups:
- Arm A (Bevacizumab): Patients receive bevacizumab 10 mg/kg IV over 30-90 minutes on days 1 and 15 in a 28-day cycle.
  bevacizumab: Given IV
- Arm B (Bevacizumab and Temsirolimus): Patients receive temsirolimus 25 mg IV over 30 minutes on days 1, 8, 15, and 22 and bevacizumab as in Arm A in a 28-day cycle.
  temsirolimus: Given IV
  bevacizumab: Given IV
- Arm C (Bevacizumab and Sorafenib): Patients receive bevacizumab 5 mg/kg IV over 30-90 minutes on days 1 and 15 and sorafenib 200 mg PO BID on days 1-5, 8-12, 15-19, and 22-26 in a 28-day cycle.
  Sorafenib: Given PO
  bevacizumab: Given IV
- Arm D (Sorafenib and Temsirolimus): Patients receive sorafenib 200 mg PO BID on days 1-28 and temsirolimus as in Arm B in a 28-day cycle.
  Sorafenib: Given PO
  temsirolimus: Given IV
Period: Overall Study
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus)
Started | 89 (Number of patients randomized to this treatment arm.) | 91 (Number of patients randomized to this treatment arm.) | 90 (Number of patients randomized to this treatment arm.) | 91 (Number of patients randomized to this treatment arm.)
Treated | 88 (Number of patients included in the toxicity analysis.) | 86 (Number of patients included in the toxicity analysis.) | 90 (Number of patients included in the toxicity analysis.) | 91 (Number of patients included in the toxicity analysis.)
Eligible and Treated | 84 (Number of patients included in the primary analysis.) | 80 (Number of patients included in the primary analysis.) | 83 (Number of patients included in the primary analysis.) | 84 (Number of patients included in the primary analysis.)
Completed | 0 (There is no limit to the number of treatment cycles allowed on any treatment arm.) | 0 (There is no limit to the number of treatment cycles allowed on any treatment arm.) | 0 (There is no limit to the number of treatment cycles allowed on any treatment arm.) | 0 (There is no limit to the number of treatment cycles allowed on any treatment arm.)
Not Completed | 89 | 91 | 90 | 91
Not completed — Disease progression | 59 | 43 | 48 | 49
Not completed — Adverse Event | 11 | 17 | 20 | 18
Not completed — Death | 2 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 4 | 8 | 5 | 7
Not completed — Physician Decision | 1 | 4 | 1 | 0
Not completed — Alternative therapy | 4 | 2 | 0 | 0
Not completed — Other complicated disease | 0 | 2 | 2 | 0
Not completed — Symptomatic deterioration | 0 | 1 | 0 | 2
Not completed — Surgery | 1 | 0 | 0 | 1
Not completed — Joint decision of physician and patient | 1 | 0 | 0 | 0
Not completed — Adverse events and progressive disease | 0 | 0 | 0 | 1
Not completed — Relocation | 0 | 0 | 1 | 0
Not completed — Ineligible | 4 | 7 | 7 | 7
Not completed — Never started treatment | 1 | 4 | 0 | 0
Not completed — Other | 1 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis.
Groups:
- Arm A (Bevacizumab): Patients receive bevacizumab 10 mg/kg IV over 30-90 minutes on days 1 and 15 in a 28-day cycle.
- Arm B (Bevacizumab and Temsirolimus): Patients receive temsirolimus 25 mg IV over 30 minutes on days 1, 8, 15, and 22 and bevacizumab as in Arm A in a 28-day cycle.
- Arm C (Bevacizumab and Sorafenib): Patients receive bevacizumab 5 mg/kg IV over 30-90 minutes on days 1 and 15 and sorafenib 200 mg PO BID on days 1-5, 8-12, 15-19, and 22-26 in a 28-day cycle.
- Arm D (Sorafenib and Temsirolimus): Patients receive sorafenib 200 mg PO BID on days 1-28 and temsirolimus as in Arm B in a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus) | Total
Number analyzed (Participants) | 84 | 80 | 83 | 84 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 51 | 52 | 61 | 213
  >=65 years | 35 | 29 | 31 | 23 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 26 | 17 | 90
  Male | 62 | 55 | 57 | 67 | 241
Region of Enrollment [Number; unit: participants]
  United States | 84 | 80 | 83 | 84 | 331

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as time from randomization to clinical evidence of disease progression or death from any cause without progression. Patients alive without progression were censored at the date of last disease assessment.
Time Frame: Assessed every 2 cycles for the first 12 cycles, then every 3 cycles until treatment discontinuation, then every 8 weeks until disease progression or up to 5 years
Population: Eligible, treated patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus)
Number analyzed (Participants) | 84 | 80 | 83 | 84
Months | 7.5 [5.8 to 10.8] | 7.6 [6.7 to 9.2] | 9.2 [7.5 to 11.4] | 7.4 [5.6 to 7.9]
Statistical Analysis 1: Comparison: Arm A (Bevacizumab) vs Arm B (Bevacizumab and Temsirolimus); Progression-free survival was compared between Arm B (bevacizumab and temsirolimus) and Arm A (bevacizumab alone) using stratified log rank test, stratified on prior cytokine or vaccine therapy and risk category (low/intermediate/high risk); Test type: Superiority or Other; p = 0.89, Log Rank
Statistical Analysis 2: Comparison: Arm A (Bevacizumab) vs Arm C (Bevacizumab and Sorafenib); Progression-free survival was compared between Arm C (bevacizumab and sorafenib) and Arm A (bevacizumab alone) using stratified log rank test, stratified on prior cytokine or vaccine therapy and risk category (low/intermediate/high risk); Test type: Superiority or Other; p = 0.54, Log Rank
Statistical Analysis 3: Comparison: Arm A (Bevacizumab) vs Arm D (Sorafenib and Temsirolimus); Progression-free survival was compared between Arm D (sorafenib and temsirolimus) and Arm A (bevacizumab alone) using stratified log rank test, stratified on prior cytokine or vaccine therapy and risk category (low/intermediate/high risk); Test type: Superiority or Other; p = 0.68, Log Rank

2. Secondary Outcome: Proportion of Patients With Stable Disease at 6 Months
Description: Patients whose date of progression was after 6 months or who were disease-free at last follow-up beyond 6 months were considered to be stable at 6 months and all other patients were not.
Time Frame: as for outcome 1
Population: Eligible, treated patients
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus)
Number analyzed (Participants) | 84 | 80 | 83 | 84
Proportion of patients | 0.548 [0.435 to 0.657] | 0.562 [0.447 to 0.673] | 0.590 [0.477 to 0.697] | 0.524 [0.412 to 0.634]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death. Patients alive at last contact were censored on the date of last contact.
Time Frame: as for outcome 1
Population: Eligible, treated patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus)
Number analyzed (Participants) | 84 | 80 | 83 | 84
Months | 28.6 [22.3 to 34.9] | 24.7 [21.4 to 35.3] | 27.5 [21.5 to 37.4] | 24.3 [19.7 to 34.7]

4. Secondary Outcome: Objective Response Rate
Description: Response was assessed using Solid Tumor Response Criteria (RECIST). Patients with complete responses or partial responses are considered having an objective response.
Time Frame: as for outcome 1
Population: Eligible, treated patients
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus)
Number analyzed (Participants) | 84 | 80 | 83 | 84
Proportion of patients | 0.133 [0.068 to 0.225] | 0.316 [0.216 to 0.431] | 0.305 [0.208 to 0.416] | 0.202 [0.123 to 0.304]
Statistical Analysis 1: Comparison: Arm A (Bevacizumab) vs Arm B (Bevacizumab and Temsirolimus); The response rate of each combination arm was compared to that of the bevacizumab alone arm; Test type: Superiority or Other; p = 0.0076, Fisher Exact — Each combination arm was compared with the bevacizumab alone arm. Since there were 3 pairwise comparisons, a Bonferroni--adjusted p-value of 0.017 was considered to be statistically significant
Statistical Analysis 2: Comparison: Arm A (Bevacizumab) vs Arm C (Bevacizumab and Sorafenib); The response rate of each combination arm was compared to that of the bevacizumab alone arm; Test type: Superiority or Other; p = 0.0085, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Arm A (Bevacizumab) vs Arm D (Sorafenib and Temsirolimus); The response rate of each combination arm was compared to that of the bevacizumab alone arm; Test type: Superiority or Other; p = 0.3006, Fisher Exact — [p-value comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Bevacizumab) | Arm B (Bevacizumab and Temsirolimus) | Arm C (Bevacizumab and Sorafenib) | Arm D (Sorafenib and Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 39/88 | 66/86 | 74/90 | 76/91
Other Adverse Events (participants affected / at risk) | 80/88 | 86/86 | 89/90 | 90/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Bevacizumab) (N=88) | Arm B (Bevacizumab and Temsirolimus) (N=86) | Arm C (Bevacizumab and Sorafenib) (N=90) | Arm D (Sorafenib and Temsirolimus) (N=91)
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 2 | 2 | 8
Leukocytes (Investigations) | 0 | 1 | 0 | 4
Lymphopenia (Investigations) | 0 | 3 | 2 | 10
Neutrophils (Investigations) | 0 | 3 | 0 | 4
Platelets (Investigations) | 0 | 2 | 1 | 8
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac-ischemia (Cardiac disorders) | 1 | 3 | 1 | 1
Cardiac troponin I (cTnI) (Investigations) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 18 | 15 | 34 | 7
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 2 | 1 | 0
Fatigue (General disorders) | 2 | 13 | 10 | 14
Fever w/o neutropenia (General disorders) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 2 | 3 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 7
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 20 | 3
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 3 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 6 | 6 | 9
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Necrosis, colon/cecum/appendix (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Obstruction, colon (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Perforation, colon (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ulcer, anus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ulcer, gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
GI-other (Gastrointestinal disorders) | 0 | 0 | 1 | 0
CNS, hemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0
Rectum, hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 0 | 1 | 0
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Infection Gr0-2 neut, abdomen (Infections and infestations) | 0 | 2 | 0 | 0
Infection Gr0-2 neut, anal/perianl (Infections and infestations) | 1 | 0 | 0 | 0
Infection Gr0-2 neut, bone (Infections and infestations) | 0 | 0 | 0 | 1
Infection Gr0-2 neut, dental-tooth (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, kidney (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 0 | 3 | 0 | 2
Infection Gr0-2 neut, rectum (Infections and infestations) | 0 | 3 | 0 | 0
Infection Gr0-2 neut, salivary (Infections and infestations) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, sinus (Infections and infestations) | 0 | 0 | 1 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 0 | 1 | 0 | 1
Infection Gr0-2 neut, wound (Infections and infestations) | 0 | 1 | 1 | 0
Infection w/ unk ANC lung (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, blood (Infections and infestations) | 0 | 1 | 0 | 0
Edema limb (General disorders) | 0 | 3 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Alkaline phosphatase (Investigations) | 0 | 1 | 0 | 1
ALT, SGPT (Investigations) | 0 | 1 | 1 | 1
Amylase (Investigations) | 0 | 0 | 2 | 4
AST, SGOT (Investigations) | 0 | 0 | 0 | 1
Bilirubin (Investigations) | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypercholesterolemia (Investigations) | 0 | 4 | 0 | 5
Creatinine (Investigations) | 0 | 1 | 3 | 0
Glomerular filtration rate (Renal and urinary disorders) | 0 | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 9 | 2 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Lipase (Investigations) | 1 | 2 | 4 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 7 | 10 | 30
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 5
Proteinuria (Renal and urinary disorders) | 9 | 22 | 9 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 8 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 5
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 1 | 2 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 3 | 6 | 4
Anus, pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Cardiac/heart, pain (Cardiac disorders) | 0 | 1 | 0 | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chest/thoracic pain NOS (General disorders) | 0 | 0 | 2 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Head/headache (Nervous system disorders) | 2 | 5 | 4 | 3
Joint, pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Neuropathic, pain (Nervous system disorders) | 0 | 1 | 0 | 0
Oral cavity, pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Rectum, pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 2
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Obstruction, airway-bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Vital capacity (Investigations) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3 | 2 | 2
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 2 | 4 | 2 | 2
Vascular-Other (Specify) (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Bevacizumab) (N=88) | Arm B (Bevacizumab and Temsirolimus) (N=86) | Arm C (Bevacizumab and Sorafenib) (N=90) | Arm D (Sorafenib and Temsirolimus) (N=91)
Allergic reaction (Immune system disorders) | 0 | 5 | 0 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 9 | 5
Hemoglobin (Blood and lymphatic system disorders) | 30 | 65 | 37 | 75
Leukocytes (Investigations) | 4 | 32 | 12 | 46
Lymphopenia (Investigations) | 7 | 21 | 16 | 28
Neutrophils (Investigations) | 2 | 21 | 3 | 22
Platelets (Investigations) | 13 | 43 | 21 | 52
Hypertension (Vascular disorders) | 29 | 39 | 42 | 34
Hypotension (Vascular disorders) | 0 | 5 | 4 | 1
Fatigue (General disorders) | 48 | 66 | 64 | 75
Fever w/o neutropenia (General disorders) | 2 | 11 | 6 | 13
Insomnia (Psychiatric disorders) | 1 | 7 | 7 | 10
Rigors/chills (General disorders) | 5 | 12 | 7 | 8
Weight loss (Investigations) | 7 | 28 | 31 | 37
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 21 | 30 | 30
Flushing (Vascular disorders) | 0 | 1 | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 10 | 13 | 14
Nail changes (Skin and subcutaneous tissue disorders) | 5 | 13 | 13 | 16
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 | 27 | 9 | 29
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 35 | 16 | 41
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 | 36 | 14 | 39
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 3 | 15 | 43 | 26
Anorexia (Metabolism and nutrition disorders) | 12 | 46 | 41 | 48
Constipation (Gastrointestinal disorders) | 14 | 24 | 23 | 24
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 15 | 40 | 45 | 65
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 2 | 6
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 5 | 7 | 19 | 7
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 | 22 | 20 | 13
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5 | 40 | 33 | 24
Nausea (Gastrointestinal disorders) | 17 | 37 | 38 | 50
Taste disturbance (Nervous system disorders) | 5 | 29 | 24 | 35
Vomiting (Gastrointestinal disorders) | 7 | 18 | 23 | 24
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 18 | 36 | 29 | 22
Infection Gr0-2 neut, sinus (Infections and infestations) | 1 | 7 | 3 | 4
Edema head and neck (General disorders) | 1 | 5 | 0 | 6
Edema limb (General disorders) | 5 | 15 | 11 | 18
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 23 | 17 | 17
Alkaline phosphatase (Investigations) | 9 | 19 | 19 | 34
ALT, SGPT (Investigations) | 11 | 23 | 11 | 36
Amylase (Investigations) | 5 | 8 | 11 | 9
AST, SGOT (Investigations) | 12 | 26 | 23 | 39
Bicarbonate (Metabolism and nutrition disorders) | 1 | 5 | 1 | 1
Bilirubin (Investigations) | 3 | 0 | 6 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 16 | 12 | 20
Hypercholesterolemia (Investigations) | 11 | 39 | 16 | 34
Creatinine (Investigations) | 25 | 43 | 37 | 35
Glomerular filtration rate (Renal and urinary disorders) | 3 | 5 | 6 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 47 | 30 | 50
Lipase (Investigations) | 7 | 13 | 23 | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 21 | 29 | 53
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 6 | 10 | 5
Hypokalemia (Metabolism and nutrition disorders) | 5 | 14 | 7 | 17
Proteinuria (Renal and urinary disorders) | 25 | 40 | 45 | 2
Hyponatremia (Metabolism and nutrition disorders) | 7 | 8 | 19 | 20
Hypertriglyceridemia (Metabolism and nutrition disorders) | 17 | 39 | 29 | 42
Metabolic/Laboratory-other (Investigations) | 2 | 10 | 10 | 8
Dizziness (Nervous system disorders) | 1 | 3 | 7 | 3
Depression (Psychiatric disorders) | 4 | 13 | 6 | 10
Neuropathy-sensory (Nervous system disorders) | 2 | 10 | 20 | 11
Tearing (Eye disorders) | 0 | 5 | 1 | 1
Abdomen, pain (Gastrointestinal disorders) | 4 | 7 | 15 | 24
Back, pain (Musculoskeletal and connective tissue disorders) | 4 | 11 | 4 | 8
Chest/thoracic pain NOS (General disorders) | 2 | 9 | 3 | 5
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 8 | 7
Head/headache (Nervous system disorders) | 13 | 28 | 23 | 22
Joint, pain (Musculoskeletal and connective tissue disorders) | 10 | 18 | 16 | 15
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 9 | 7
Oral cavity, pain (Gastrointestinal disorders) | 0 | 6 | 4 | 4
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 22 | 9 | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 30 | 13 | 21
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 0 | 4
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 30 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less